CLINICAL TRIAL: NCT01433224
Title: Genomic Signatures of Malignant Germ Cell Tumor Progression: A Retrospective Study of Banked Specimens
Brief Title: Studying Biomarkers in Samples From Younger Patients With Malignant Germ Cell Tumor Progression
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AGCT11B2; COG-AGCT11B2 (Other: Children's Oncology Group); AGCT11B2 (Other: Children's Oncology Group); NCI-2011-03456 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: recurrent childhood malignant germ cell tumor; recurrent extragonadal germ cell tumor; recurrent malignant testicular germ cell tumor; recurrent ovarian germ cell tumor
MeSH Terms: conditions — Ovarian Neoplasms; Testicular Germ Cell Tumor; Testicular Neoplasms | interventions — DNA Methylation; Base Sequence; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: RNA analysis
Genetic: mutation analysis
Genetic: nucleic acid sequencing
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors find better ways to treat cancer.

PURPOSE: This research trial studies samples from younger patients with malignant germ cell tumor progression.

DETAILED DESCRIPTION:
OBJECTIVES:

* Explore inter-tumoral heterogeneity in DNA methylation by tumor histology.
* Determine the genomic methylation pattern in the tumors.
* Correlate methylation pattern with tumor histology and clinical characteristics.
* Carry out exome capture and massively parallel sequencing on selected germ cell tumors (GCTs) and matched normal tissue.
* Perform exome capture and Solexa sequencing on a selected set of GCTs.
* Validate candidate mutations in an independent set of tumors.
* Determine the expression profile of mRNAs, lincRNAs and microRNAs in the tumors using RNA Seq.

OUTLINE: Archived blood and tumor tissue samples are analyzed for genomic methylation pattern, exome capture and sequencing, and candidate mutations by methylation-specific PCR techniques, single nucleotide polymorphism (SNP) arrays, and Solexa sequencing methods. Results are validated by using pyrosequencing assays and primer-extension assays. Methylation pattern is also associated with each patient's tumor histology and clinical data.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Tumor and blood specimens from patients registered on the Children Oncology Group (COG) Germ Cell Tumor Protocols, and from other study sites for non-COG patients, including Children's Medical Center, Dallas and the Dana-Farber Cancer Institute, Boston
* Patients' clinical data

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients registered on the Children Oncology Group (COG) Germ Cell Tumor Protocols.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2011-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Event-free survival
Genomic prognostic signatures associated with GCTS
Genetic variants that contribute to GCTS pathogenesis
Expression of various forms of RNA

CONTACTS AND LOCATIONS:
Overall Officials: James F. Amatruda, MD, PhD, Principal Investigator — Simmons Cancer Center